CLINICAL TRIAL: NCT02637856
Title: An Open-Label Study to Evaluate the Effectiveness and Safety of Ocrelizumab in Patients With Relapsing Remitting Multiple Sclerosis Who Have Had a Suboptimal Response to an Adequate Course of Disease-Modifying Treatment
Brief Title: A Study of Ocrelizumab in Participants With Relapsing Remitting Multiple Sclerosis (RRMS) Who Have Had a Suboptimal Response to an Adequate Course of Disease-Modifying Treatment (DMT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MN30035
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ocrelizumab (Experimental): Participants will receive ocrelizumab as an initial dose of two 300-mg IV infusions (600 mg total) separated by 14 days (on Days 1 and 15) followed by one 600-mg IV infusion every 24 weeks for a maximum of 4 doses (up to 96 weeks).
  Interventions: Drug: Ocrelizumab
- Ocrelizumab (substudy) (Experimental): Participants with no serious IRR throughout the main study will be eligible to enroll in an optional substudy and receive one additional shorter infusion of ocrelizumab at the Week 96 visit. Ocrelizumab will be administered IV as a single 600-mg dose at a shorter infusion rate (approximately 2 hours instead of 3.5 hours)
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Participants will receive ocrelizumab as an initial dose of two 300-mg IV infusions (600 mg total) separated by 14 days (on Days 1 and 15) followed by one 600-mg IV infusion every 24 weeks for a maximum of 4 doses (up to 96 weeks).
  Other Names: RO4964913
  Arms: Ocrelizumab
Drug: Ocrelizumab — Participants will receive an additional single 600-mg dose IV infusion at a shorter infusion rate (approximately 2 hours instead of 3.5 hours)
  Other Names: RO4964913
  Arms: Ocrelizumab (substudy)

SUMMARY:
This study will evaluate the efficacy and safety of ocrelizumab in participants with RRMS who have had a suboptimal response to an adequate course of DMT. Participants will receive ocrelizumab as an initial dose of two 300-milligrams (mg) intravenous (IV) infusions (600 mg total) separated by 14 days followed by one 600-mg IV infusion for a maximum of 4 doses (up to 96 weeks). Anticipated time on study treatment is 96 weeks.

DETAILED DESCRIPTION:
Participants who complete their Week 72 ocrelizumab infusion and do not experience any serious infusion related reaction (IRR) throughout the main study will be eligible to enroll in an optional, open-label, non-randomized substudy to MN30035 and receive one additional shorter infusion of ocrelizumab at the Week 96 visit. This substudy will enroll approximately 100 patients from MN30035 main study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis (specifically RRMS), in accordance with the revised 2010 McDonald criteria
* Disease duration from first symptom of less than or equal to (</=) 12 years
* Treated with an adequate course of treatment with no more than three prior DMT regimens of greater than or equal to (>/=) 6 months, and the discontinuation of the most recent adequately used DMT was due to suboptimal response
* Suboptimal response while the participant was on his/her last adequately used DMT for >/=6 months (defined by having one of the following qualifying events despite being on a stable dose of the same DMT for at least 6 months: one or more clinically reported relapses, one or more T1 Gd-enhanced lesions, or two or more new or enlarging T2 lesions on MRI); these qualifying events must have occurred while on the last adequately used DMT. In participants receiving stable doses of the same approved DMT for more than a year, the event must have occurred within the last 12 months of treatment with this DMT from the date of screening

Exclusion Criteria:

* History of primary progressive multiple sclerosis (PPMS), progressive relapsing multiple sclerosis (PRMS), or secondary progressive multiple sclerosis (SPMS)
* Contraindications for MRI
* Known presence of other neurological disorders that may mimic multiple sclerosis
* Pregnancy or lactation, or intention to become pregnant during the study
* Requirement for chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* History of or currently active primary or secondary immunodeficiency
* Lack of peripheral venous access
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Active infection, or history of or known presence of recurrent or chronic infection such as human immunodeficiency virus (HIV), syphilis, or tuberculosis
* History of progressive multifocal leukoencephalopathy
* Contraindications to or intolerance of oral or IV corticosteroids
* Previous treatment with fingolimod (Gilenya®) or dimethyl fumarate (Tecfidera®) in participants whose lymphocyte count is below the lower limit of normal (LLN)
* Treatment with alemtuzumab (Lemtrada®)
* Previous treatment with systemic cyclophosphamide, azathioprine, mycophenolate mofetil, cyclosporine, or methotrexate
* Previous treatment with natalizumab within 12 months prior to screening unless failure was due to confirmed, persistent anti-drug antibodies (ADAs). Participants previously treated with natalizumab will be eligible for this study only if duration of treatment with natalizumab was less than (<) 1 year and natalizumab was not used in the 12 months prior to screening. Anti-John Cunningham virus (JCV) antibody status (positive or negative) and titer (both assessed within the year of screening) must be documented prior to enrollment
* Treatment with dalfampridine (Ampyra®) unless on stable dose for >/=30 days prior to screening
* Treatment with a B-cell targeted therapies (e.g., rituximab, ocrelizumab, atacicept, belimumab, or ofatumumab)
* Treatment with a drug that is experimental (Exception: treatment with an experimental drug that was subsequently approved in the participant's country is allowed)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 608 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (82):
- United States (67):
  - North Central Neurology Associates, Cullman, Alabama
  - Phoenix Neurological Associates Ltd, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Territory Neurology and Research Institute, Tucson, Arizona
  - The Research Center of Southern California, LLC, Carlsbad, California
  - Mercy Medical Group; MS Centre Nurse, Carmichael, California
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Scripps Health, La Jolla, California
  - UCSF- Multiple Sclerosis Centre; Department of Neurology, San Francisco, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Mountain Neurological Research Center; Roaring Fork Neurologt, P.C., Basalt, Colorado
  - IMMUNOe Research Centers, Centennial, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - Advanced Neurology of Colorado, LLC, Fort Collins, Colorado
  - Associated Neurologists of Southern CT PC, Fairfield, Connecticut
  - KI Health Partners, LLC; New England Institute for Clinical Research, Stamford, Connecticut
  - Neurology Associates PA, Maitland, Florida
  - University of Miami Miller School of Medicine; Clinical Reseach Building, Miami, Florida
  - Neurostudies Inc, Port Charlotte, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University of South Florida - Bradenton, Tampa, Florida
  - Ms Center Of Atlanta, Atlanta, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - Consultants in Neurology Ltd, Northbrook, Illinois
  - American Health Network Institute, LLC, Avon, Indiana
  - Josephson Wallack Munshower Neurology PC, Indianapolis, Indiana
  - University of Kansas Medical Center; Division of Nuclear Medicine, Kansas City, Kansas
  - Lahey Clinic Med Ctr, Lexington, Kentucky
  - Associates in Neurology PSC, Lexington, Kentucky
  - Community Medical Associates Inc.; d.b.a. Norton Neurology Services MS Services, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Medical Center; Department of Neurology, Baltimore, Maryland
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr; Neurology/MS Center, Boston, Massachusetts
  - Dragonfly Research, LLC, Wellesley, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Wayne State University; Department of Neurology, Detroit, Michigan
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Washington University School of Medicine; Department of Neurology, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo; Center for Brain Research, Las Vegas, Nevada
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Holy Name Hospital; Institute For Clinical Research, Teaneck, New Jersey
  - Jacobs Neurological Institute, Buffalo, New York
  - The MS Center of Northeastern New York, Latham, New York
  - Columbia University Medical Center, New York, New York
  - South Shore Neurologic Associates P.C., Patchogue, New York
  - Island Neurological Associates, P.C., Plainview, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - Cleveland Clinic Foundation; Cleveland Clinic Cancer Center/I40, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center; Department of Neurology, Columbus, Ohio
  - Neurology Specialists, Inc, Dayton, Ohio
  - Neurology and Neuroscience Assoc., Inc., Westerville, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Providence Multiple Sclerosis Center, Portland, Oregon
  - Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - Neurology Clinic PC, Cordova, Tennessee
  - Hope Neurology, Knoxville, Tennessee
  - Uni of Texas Health Science Center At Houston, Houston, Texas
  - Bhupesh Dihenia M.D. P.A., Lubbock, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
  - Rocky Mountain MS Clinic, Salt Lake City, Utah
  - Swedish Neuroscience Institute, Seattle, Washington
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
- Canada (15):
  - Foothills Medical Centre; Centre Dept of Medical Clinical Neuroscience, Calgary, Alberta
  - University of Alberta; Divison of Pulmonary Medicine, Dept. of Medicine,, Edmonton, Alberta
  - Fraser Health Multiple Sclerosis Clinic; Burnaby Hospital Pharmacy, Burnaby, British Columbia
  - Horizon Health Network - Multiple Sclerosis Clinic, Saint John, New Brunswick
  - Dalhousie Multiple Sclerosis Research Unit, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - The Ottawa Hospital - General Campus; Department of Neurology - Multiple Sclerosis, Ottawa, Ontario
  - St. Michael's Hospital MS Clinic, MS Research Centre, Toronto, Ontario
  - Clinique NeuroOutaouais, Gatineau, Quebec
  - Recherche Sepmus, Inc., Greenfield Park, Quebec
  - Hopital Hotel Dieu de Levis, Lévis, Quebec
  - Chum Campus Notre Dame, Montreal, Quebec
  - McGill University; Montreal Neurological Institute; Neurological and Psychiatric, Montreal, Quebec
  - MS Clinic Mauricie Bois Francs, Trois-Rivières, Quebec
  - CHU De Quebec Universite Laval, Québec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in North America at 90 study sites in the U.S. and Canada.
Pre-assignment Details: Participants with relapsing remitting multiple sclerosis (RRMS) were enrolled, who had had a suboptimal response to an adequate course of a disease-modifying treatment (DMT). An adequate course of prior DMT was defined as the same DMT administered for at least 6 months.
Groups:
- Ocrelizumab: Participants received ocrelizumab as an initial dose of two 300-mg IV infusions (600 mg total) separated by 14 days (on Days 1 and 15) followed by one 600-mg IV infusion every 24 weeks for a maximum of 4 doses (up to 96 weeks)
- Ocrelizumab (Substudy): Participants who completed their Week 72 ocrelizumab infusion and did not experience any serious infusion related reactions (IRRs) throughout the main study were eligible to enroll in an optional substudy and received one additional shorter infusion of ocrelizumab at the Week 96 visit. Ocrelizumab was administered as a single 600-mg dose at a shorter infusion rate (approximately 2 hours instead of 3.5 hours)
Period: Main Study (Baseline to Week 100)
Arm/Group | Ocrelizumab | Ocrelizumab (Substudy)
Started | 608 | 0
Completed | 389 | 0
Not Completed | 219 | 0
Not completed — Adverse Event | 9 | 0
Not completed — Lost to Follow-up | 5 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Pregnancy | 7 | 0
Not completed — Withdrawal by Subject | 20 | 0
Not completed — Protocol Deviation | 2 | 0
Not completed — Continued on Commercial Ocrevus | 164 | 0
Not completed — Failed Drug Test | 1 | 0
Not completed — Incarceration | 1 | 0
Not completed — Pregnancy Attempts | 2 | 0
Not completed — Site Closing | 6 | 0
Period: Sub-Study (Week 72 to Week 100)
Arm/Group | Ocrelizumab | Ocrelizumab (Substudy)
Started | 0 | 129
Completed | 0 | 125
Not Completed | 0 | 4
Not completed — Non-safety reason (moved out of state) | 0 | 1
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 438
  Male | 170
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 68
  Not Hispanic or Latino | 526
  Not Stated | 7
  Unknown | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 13
  Black or African American | 72
  Multiple | 6
  Native Hawaiian or other Pacific Islande | 3
  Unknown | 17
  White | 495

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Any Protocol-Defined Events During 96-Week Period
Description: Protocol-defined event is the occurrence of either protocol-defined relapse (occurrence of new or worsening neurological symptoms attributable to multiple sclerosis) or T1 gadolinium (Gd)-enhanced lesion on brain magnetic resonance imaging (MRI) or new and/or enlarging T2 lesion on brain MRI or confirmed disability progression at 24 weeks.
Time Frame: Baseline up to Week 96
Population: The modified Intent-to-Treat (mITT) population was a subset of the ITT population which excluded participants who discontinued ocrelizumab treatment early without any protocol-defined events for reasons other than death and lack of efficacy. Only participants for whom data were collected are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Percentage of Participants | 48.1 [43.9 to 52.3]

2. Secondary Outcome: Percentage of Participants Without Any Protocol-Defined Events During 24-Week and 48-Week Period
Description: Protocol-defined event is the occurrence of either protocol-defined relapse (occurrence of new or worsening neurological symptoms attributable to multiple sclerosis) or T1 Gd-enhanced lesion on brain MRI or new and/or enlarging T2 lesion on brain MRI or confirmed disability progression at 24 weeks.
Time Frame: Baseline up to Weeks 24 and 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Percentage of Participants
  Week 24: number analyzed (Participants) | 576
  Week 24 | 59.0 [54.9 to 63.1]
  Week 48: number analyzed (Participants) | 576
  Week 48 | 51.2 [47.0 to 55.4]

3. Secondary Outcome: Time to Protocol-Defined Event
Description: as for outcome 2
Time Frame: Baseline up to Week 96
Population: All enrolled participants who received any ocrelizumab. Participants who prematurely withdrew from the study for any reason and who did not have any assessments for any reason were still included in the ITT population as long as the participant received ocrelizumab
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Weeks | NA [53.86 to NA] — Not estimable because more than 50% of the ITT population were event-free at the end of the study

4. Secondary Outcome: Total Number of Protocol-Defined Relapses Per Participant Year During 96-week Period
Description: Protocol-defined relapse is an occurrence of new or worsening neurological symptoms attributable to multiple sclerosis which must persist for greater than (>) 24 hours and should not be attributable to confounding clinical factors (e.g., fever, infection, injury, adverse reactions to medications) and immediately preceded by a stable or improving neurological state for least 30 days. The Adjusted Annualized Relapse Rate was adjusted by baseline Expanded Disability Status Scale (EDSS <2.5 vs. >=2.5) and number of previous disease-modifying treatments (DMTs =1 vs. >1)
Time Frame: Baseline up to Week 96
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Number of Relapses/Participant Year
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Number of Relapses/Participant Year | 0.046 [0.036 to 0.060]

5. Secondary Outcome: Time to Onset of First Protocol-Defined Relapse
Description: Protocol-defined relapse is an occurrence of new or worsening neurological symptoms attributable to multiple sclerosis which must persist for >24 hours and should not be attributable to confounding clinical factors (e.g., fever, infection, injury, adverse reactions to medications) and immediately preceded by a stable or improving neurological state for least 30 days.
Time Frame: Baseline up to Week 96
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Weeks | NA [NA to NA] — Not estimable because more than 50% of the ITT population were event-free at the end of the study

6. Secondary Outcome: Time to Onset of First T1 Gd-Enhanced Lesion as Detected by Brain MRI
Time Frame: Baseline up to Week 96
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Weeks | NA [NA to NA] — Not estimable because more than 50% of the ITT population were event-free at the end of the study

7. Secondary Outcome: Time to Onset of First New and/or Enlarging T2 Lesion as Detected by Brain MRI
Time Frame: Baseline up to Week 96
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Weeks | NA [NA to NA] — Not estimable because more than 50% of the ITT population were event-free at the end of the study

8. Secondary Outcome: Time to Onset of Confirmed Disability Progression (CDP) for at Least 24 Weeks According to Expanded Disability Status Scale (EDSS) Score
Time Frame: Baseline up to Week 96
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Weeks | NA [NA to NA] — Not estimable because more than 50% of the ITT population were event-free at the end of the study

9. Secondary Outcome: Total Number of T1 Gd-Enhancing Lesions as Detected by Brain MRI
Description: The analyses included participants who had an interpretable MRI at the time point of interest. Participants having 0, 1, 2, 3, and greater than 3 lesions at weeks 24, 48, and 96 were included in the analysis.
Time Frame: Weeks 24, 48, and 96
Population: All enrolled participants who received any ocrelizumab. Participants who prematurely withdrew from the study for any reason and who did not have any assessments for any reason were still included in the ITT population as long as the participant received ocrelizumab. Only participants for whom data were collected are included in the analysis.
Measure: Number; unit: Number of Lesions
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Number of Lesions
  Week 24: number analyzed (Participants) | 599
  Week 24 | 33 [0.010 to 0.050]
  Week 48: number analyzed (Participants) | 582
  Week 48 | 16 [0.002 to 0.031]
  Week 96: number analyzed (Participants) | 557
  Week 96 | 7 [0.002 to 0.026]

10. Secondary Outcome: Change From Baseline in Total T2 Lesion Volume as Detected by Brain MRI
Description: Baseline data is represented as mean; post-Baseline date are represented as mean changes.
Time Frame: Baseline, Weeks 24, 48, and 96
Population: as for outcome 9
Measure: Mean (Standard Error); unit: cubic centimeter (cm3)
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
cubic centimeter (cm3)
  Baseline: number analyzed (Participants) | 600
  Baseline | 11.551 (0.590)
  Week 24: number analyzed (Participants) | 595
  Week 24 | -0.484 (0.118)
  Week 48: number analyzed (Participants) | 579
  Week 48 | -0.549 (0.123)
  Week 96: number analyzed (Participants) | 554
  Week 96 | -0.560 (0.129)

11. Secondary Outcome: Total Number of New and/or Enlarging T2 Lesions as Detected by Brain MRI
Time Frame: Weeks 24, 48, and 96
Population: as for outcome 9
Measure: Number; unit: Number of Lesions
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Number of Lesions
  Week 24: number analyzed (Participants) | 598
  Week 24 | 640
  Week 48: number analyzed (Participants) | 583
  Week 48 | 39
  Week 96: number analyzed (Participants) | 558
  Week 96 | 38

12. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to 100 weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 608
Percentage of Participants | 86.3

13. Primary Outcome: Percentage of Participants With Infusion Related Reactions (IRRs) in Optional Substudy
Description: Rate and frequency of Grade 3 or 4 IRRs with onset on or after the shorter ocrelizumab infusion
Time Frame: Week 96 to Week 100
Population: Participants who completed their Week 72 ocrelizumab infusion and did not experience any serious IRRs throughout the main study
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab (Substudy)
Number analyzed (Participants) | 129
Percentage of Participants | 0 [0.0 to 2.8]

ADVERSE EVENTS:
Time Frame: Baseline up to 100 weeks
Description: The Safety Population included all enrolled participants who received any ocrelizumab.
Arm/Group | Ocrelizumab | Ocrelizumab (Substudy)
All-Cause Mortality (participants affected / at risk) | 0/608 | 0/129
Serious Adverse Events (participants affected / at risk) | 47/608 | 2/129
Other Adverse Events (participants affected / at risk) | 406/608 | 16/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab (N=608) | Ocrelizumab (Substudy) (N=129)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (2) | 0 (0)
Mastoid effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 3 (3) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (3) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Fibromuscular dysplasia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab (N=608) | Ocrelizumab (Substudy) (N=129)
Nausea (Gastrointestinal disorders) | 32 (38) | 0 (0)
Fatigue (General disorders) | 58 (62) | 0 (0)
Nasopharyngitis (Infections and infestations) | 64 (81) | 0 (0)
Sinusitis (Infections and infestations) | 37 (47) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 57 (76) | 0 (0)
Urinary tract infection (Infections and infestations) | 88 (118) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 263 (519) | 16 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36 (41) | 0 (0)
Headache (Nervous system disorders) | 56 (66) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT02637856/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT02637856/SAP_001.pdf